CLINICAL TRIAL: NCT01289288
Title: A Physician-Based Trial to Increase Colorectal Cancer Screening in Chinese
Acronym: CRC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Temple University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Judy Wang, Assistant Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007-297; R01CA121023 (NIH)
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer screening; Chinese Americans; patients nonadherent with CRC Screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mailed printed materials and in-office training (Experimental)
  Interventions: Behavioral: Mailed printed materials and in-office training
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Mailed printed materials and in-office training — 1. Mailed printed materials including CRC physician guide, patient brochure, flip chart and a poster
  2. Two sessions of in-office training with two standardized patients
  Arms: Mailed printed materials and in-office training

SUMMARY:
The objective of this study is to test whether a culturally-tailored in-office based intervention have impact on increasing Chinese physician's recommendation of colorectal cancer (CRC) screening to their nonadherent Chinese patients.

Special aims are to:

1. Evaluate the efficacy of a culturally-tailored physician intervention on increasing non-adherent Chinese American's patients' CRC screening rate.
2. Identify factors that mediate or moderate the intervention effects. For example, patients who hold an eastern cultural view or are less acculturated will be more likely to benefit from the intervention than patients who hold a western view or who are more acculturated.

DETAILED DESCRIPTION:
This study is a randomized controlled trial aiming to test the effect of the culturally-tailored in-office based intervention on physicians. A total of 24 Chinese physicians in the Washington DC and Philadelphia areas and a total of 24 eligible Chinese patients from each physician will be recruited for this study. Physicians and their patients are randomized into two groups: A and B. Physician in the intervention group (A) will receive mailed printed materials including a CRC physician guide, patient brochure, flip chart and a poster and two sessions of in-office training aimed to reinforce learning of the topic covered by the mailed materials and provide physicians with hands-on experience in using communication skills with standardized patients. Physicians in the control group (B) will receive nothing until the end of the study. Patients will be followed 12-month later after their completion of the baseline survey and their self-reported CRC screening status will be verified by chart audit.

ELIGIBILITY:
Inclusion Criteria:

For Physicians

1. are Chinese American,
2. practice primary care,
3. have a least 75 Chinese patients aged 50 and older in their practice,
4. can communicate with patients in Chinese (Mandarin, Cantonese, etc.)

For Patients

1. visiting the participating physician at least once in the past 2 years,
2. are Chinese Americans,
3. are 50 years and older,
4. never had any CRC screening or are overdue for screening.

Exclusion Criteria:

For Patients:

1. have a colorectal polyp, CRC cancer, or a family history of CRC (first degree relative), and
2. had updated CRC screening (FOBT within one year, colonoscopy within 10 years, sigmoidoscopy within 5 years and double-contrast barium enema within 5 years).

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2007-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Receipt of CRC screening | 12 months
  Nonadherent Chinese American patient's CRC screening rates.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Wang, Ph.D., Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Georgetown University, Washington D.C., District of Columbia
  - Temple University, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Liang W, Wang JH, Chen MY, Mandelblatt JS. Language use and the receipt of cancer screening recommendations by immigrant Chinese American women. J Womens Health (Larchmt). 2009 Feb;18(2):201-7. doi: 10.1089/jwh.2007.0709. PMID 19183091
- [Background] Wang JH, Liang W, Chen MY, Cullen J, Feng S, Yi B, Schwartz MD, Mandelblatt JS. The influence of culture and cancer worry on colon cancer screening among older Chinese-American women. Ethn Dis. 2006 Spring;16(2):404-11. PMID 17682242
- [Derived] Huei-Yu Wang J, Ma GX, Liang W, Tan Y, Makambi KH, Dong R, Vernon SW, Tu SP, Mandelblatt JS. Physician Intervention and Chinese Americans' Colorectal Cancer Screening. Am J Health Behav. 2018 Jan 1;42(1):13-26. doi: 10.5993/AJHB.42.1.2. PMID 29320335
- [Derived] Wang JH, Sheppard VB, Liang W, Ma GX, Maxwell AE. Recruiting Chinese Americans into cancer screening intervention trials: strategies and outcomes. Clin Trials. 2014 Apr;11(2):167-77. doi: 10.1177/1740774513518849. Epub 2014 Feb 24. PMID 24567288